CLINICAL TRIAL: NCT00718250
Title: A Phase I Study of Lentivirus Transduced Acute Myeloid Leukaemic Cells (AML) Expressing B7.1 (CD80) and IL-2 for the Potential Enhancement of Graft Versus Leukaemia(GvL) Effect in Poor Prognosis AML
Brief Title: Lentivirus Transduced Acute Myeloid Leukaemia Blasts Expressing B7.1 (CD80) and IL-2
Acronym: RFUSIN2-AML1
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Collaborators: Department of Health (Ambiguous); Leukemia Research Fund (Other); Elimination of Leukaemia Fund (Other)
Responsible Party: Dr Lorraine Catt, Research and Development Manager, King's College Hospital NHS Foundation Trust, London, United Kingdom
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: O5CC14; EudraCT 2005-000806-29; GTAC GTAC098
Record Dates: First submitted 2008-06-06; First posted 2008-07-18 (Estimated); Last update posted 2008-07-18 (Estimated); Status verified 2008-07

CONDITIONS: Leukemia, Myeloid, Acute
Keywords: Acute myeloid leukaemia; Cancer vaccines; Immunotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- cohort 1 (Experimental): AML Cell Vaccine alone
  Interventions: Biological: RFUSIN2-AML1
- cohort 2 (Experimental): Donor leukocytes alone
  Interventions: Biological: Donor leukocyte infusion (DLI)
- cohort 3 (Experimental): AML cell vaccine and Donor Leukocyte Infusion (1x107/kg)
  Interventions: Biological: RFUSIN2-AML1 and donor leukocyte infusion
- cohort 4 (Experimental): AML cell vaccine and Donor Leukocyte Infusion (1x108/kg)
  Interventions: Biological: RFUSIN2-AML1 and donor leukocyte infusion

INTERVENTIONS:
Biological: RFUSIN2-AML1 — AML cell vaccine alone. x4 doses 3 weeks apart
  Arms: cohort 1
Biological: Donor leukocyte infusion (DLI) — 1 dose 1x107/kg
  Other Names: RFUSIN2-AML1
  Arms: cohort 2
Biological: RFUSIN2-AML1 and donor leukocyte infusion — AML cell vaccine x 4 doses 3 weeks apart Donor leukocyte infusion 1x107/kg x 1 dose
  Other Names: RFUSIN2-AML1
  Arms: cohort 3
Biological: RFUSIN2-AML1 and donor leukocyte infusion — AML cell vaccine x4 doses 3 weeks apart Donor leukocyte infusion 1x108/kg x1 dose
  Other Names: RFUSIN2-AML1
  Arms: cohort 4

SUMMARY:
The purpose of this study is to assess the safety and tolerability of an 'AML Cell Vaccine' in patients with poor prognosis acute myeloid leukaemia (AML).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AML defined according to the WHO classification
* Age ≥ 18 years
* New presentation or relapsed AML
* Patients must be able to give written informed consent
* Failure to enter complete morphological remission (>5% bone marrow AML cells) or persistence of cytogenetic abnormality following intensive combination chemotherapy At day+100 post-transplant
* HIV negative
* No GvHD
* No continuing use of immunosuppressive drugs
* Absence of active systemic fungal or viral infection including HTLV-1, hepatitis B or C.
* Adequate renal and liver function confirmed by: creatinine clearance >30mls/min; bilirubin <3.0 x upper limit of normal; AST <3.0 x upper limit of normal; prothrombin time <2.0 x upper limit of normal.

Performance status of 1 or less by ECOG criteria or >80% by the Karnovsky score

* Patient must provide written informed consent and be willing to comply for the duration of the study.
* Life expectancy >36 weeks
* Women of childbearing potential (WCBP) must have a negative serum or urine pregnancy test within 10 - 14 days and again within 24 hours of starting the study. In addition, sexually active WCBP must agree continued abstinence from heterosexual intercourse or to use adequate contraceptive methods starting 4 weeks prior to the initiation of therapy (see appendix G for pregnancy testing and birth control guidelines while on study). WCBP must agree to have pregnancy tests every 3 weeks while on study drug (every 14 days for women with irregular cycles) and 4 weeks after the last dose of study drug. Men must also agree to use a condom if their partner is of child bearing potential, even if they have had a successful vasectomy.

Exclusion Criteria:

* Age < 18 years
* Patients not fit for intensive chemotherapy
* Complete morphological and cytogenetic remission following intensive combination chemotherapy
* Absence of HLA compatible donor
* HIV positive
* Evidence of graft versus host disease at day+100 post transplant
* Evidence of relapse of leukaemia (≥5% bone marrow blasts)
* Concurrent use of other forms of anti-leukaemic therapy
* Other malignancy with the exception of carcinoma in situ.
* Significant history of heart disease (unstable angina, myocardial within the past six months, congestive cardiac failure requiring daily treatment)
* Evidence of active lung disease determined by chest x-ray and absence of chronic lung disease (FEV1<60% predicted, Vital capacity <60%, Tlco<50%)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2008-05; Primary Completion 2011-05 (Estimated); Study Completion 2012-02 (Estimated)

PRIMARY OUTCOMES:
Toxicity and safety of the 'AML Cell Vaccine' | one year

SECONDARY OUTCOMES:
relapse, leukaemia free survival and overall survival | one year

CONTACTS AND LOCATIONS:
Overall Officials: Ghulam J Mufti, Principal Investigator — King's College London, London, United Kingdom
Locations (1):
- King's College Hospital NHS Foundation Trust, London, London, United Kingdom